CLINICAL TRIAL: NCT05616338
Title: Modeling Bronchial Epithelium in Severe Asthma With Human Induced Pluripotent Stem Cells (iPSC)
Acronym: MOSAIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0384; 2022-A02059-34 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2023-08

CONDITIONS: Severe Asthma; Allergic Bronchopulmonary Aspergillosis (ABPA)
Keywords: Severe asthma; ABPA; Pluripotent stem cells; Airway epithelium; Eosinophils; Crystal
MeSH Terms: conditions — Asthma; Aspergillosis, Allergic Bronchopulmonary | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eligible patients (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A blood sample and a nasal brush for each participant. The nasal brushing will allow the isolation of epithelial cells that will serve as a comparison for the bronchial tissue produced from blood-derived iPS.
  A blood sample of approximately 14 ml will be taken for isolation and freezing of the blood mononuclear cells allowing the generation of iPS.
  Other Names: nasal brush

SUMMARY:
Asthma is severe when it cannot be controlled with maximum-dose inhaled therapies while management of comorbidities and other precipitating or aggravating factors has been optimized. Allergic bronchopulmonary aspergillosis (ABPA) is a complex bronchopulmonary disease resulting from immunological reactions against Aspergillus Fumigatus.

The development of a model of bronchial epithelium generated from patients with chronic lung disease will allow the modeling of bronchial tissue to understand the formation of these mucus plugs. This study aims to validate this model

The investigators propose to verify the feasibility of obtaining and comparing two epithelia in two populations based on the following experiments:

Differentiation of an Induced Pluripotent Stem cell (iPSC) clone derived from blood sample (Peripheral Blood Mononuclear Cells) of Type 2 inflammation (T2) severe asthma and Allergic Bronchopulmonary Aspergillosis (ABPA) in order to obtain differentiated bronchial epithelia in vitro.

DETAILED DESCRIPTION:
Asthma is severe when it cannot be controlled with maximum-dose inhaled therapies while management of comorbidities and other precipitating or aggravating factors has been optimized. Allergic bronchopulmonary aspergillosis (ABPA) is a complex bronchopulmonary disease resulting from immunological reactions against Aspergillus Fumigatus.

At the cellular and molecular level, severe asthma and ABPA are chronic bronchial diseases characterized by type 2 (T2) airway inflammation, bronchial smooth muscle hyperplasia, excessive mucus production by mucus cell metaplasia and epithelial remodeling. Type 2 inflammation in asthma is predominant and is characterized by the accumulation of immune cells, such as eosinophils, mast cells, T-helper 2 (Th2) cells, innate lymphoid cells type 2 (ILC2s) and dendritic cells.

Persistent airway obstruction despite maximal therapy is currently considered the greatest unmet medical need in asthma treatment. Fahy and colleagues published a key paper in 2018 that may explain airway obstruction. Using chest CT scans, they demonstrated the presence of mucus plugs that completely occlude segments of the airways of severe asthmatics. These mucus plugs are associated with a high number of circulating eosinophils in the blood.

There is no large-scale model to model severe asthma and ABPA. The investigators propose to develop a bronchial epithelium with pluripotent stem cells (iPSC) in air-liquid interface called iALI generated from these patients in aim to model severe asthma and ABPA and in particular the epithelium.

The secondary objectives aims to answer are:

* Comparison of the iPSC derived airway epithelium with nasal epithelial cells isolated from the same patient (nasal brush).
* To characterize the phenotype of the iPSC derived airway epithelium from ABPA and T2 severe asthma patient, in comparison to a healthy control.
* Differentiation of iPSC into mature eosinophils
* Co culture of the epithelia with iPSC derived eosinophils
* Culture of iPSC derived airway epithelium with Charcot-Leyden crystal
* Demonstrate the feasibility of obtaining iPSC from peripheral blood sampling.

ELIGIBILITY:
Inclusion Criteria:

- Smoking < 10 BP and weaned > 1 year.

Diagnostic criteria for Severe asthma group T2 :

* History of severe asthma diagnosed by a physician (according to GINA criteria)
* Subject on high dose inhaled corticosteroid (ICS 1000 µg beclometasone equivalent) and beta-agonists for at least 6 months prior to inclusion
* Blood eosinophilia in history (previous years) > 300/mm3

Diagnostic criteria for Allergic bronchopulmonary aspergillosis (ABPA) group

- Diagnosis of ABPA defined by the following 3 mandatory criteria:

1. Diagnosis of asthma by the physician for at least 12 months based on the 2019 recommendations of the Global Initiative for Asthma (GINA) group
2. Evidence of hypersensitivity to Aspergillus Fumigatus by skin test (on screening or previous documented positive skin test within the last 12 months), or serum Immunoglobulin E (IgE) specific antibodies to A. Fumigatus (≥ 0.35 kUnit/l) at screening.
3. Elevated total serum IgE (> 1000 IU/ml). If the 3 ancillary criteria for the diagnosis of of ABPA (below) are met, an IgE level ≤ 1,000 IU/ml is acceptable. If the patient is receiving oral corticosteroids (OCs) at screening, a previous documented IgE level >1000 IU/ml within the last 12 months is acceptable.

And at least 2 of the following ancillary criteria:

1. Blood eosinophil count >500 cells/μl at screening for patients not receiving OCs at screening. For patients receiving OCs at screening, blood eosinophil count > 500 cells/μl at screening or documented previous eosinophil count > 500 cells/μl in the last 12 months.
2. Presence of precipitating antibodies or serum immunoglobulin G (IgG) to A. Fumigatus at screening.
3. Documented radiological abnormalities consistent with ABPA (such as transient mucoid impaction, hyperdense mucus [high attenuation of mucous plugs], opacities of centro-lobular nodules attenuation of mucous plugs], opacities of centro-lobular nodules, telectasis, bronchiectasis, etc.) by chest X-ray or high-resolution computed tomography (HR-CT) within the last 18 months or at screening.

Exclusion Criteria:

* Other associated respiratory diseases (e.g. chronic obstructive pulmonary disease (COPD), cystic fibrosis)
* Patient in an exclusion period determined by another protocol
* Protected populations according to the French public health code: Parturient, nursing or pregnant women; subjects deprived of liberty by judicial or administrative decision; Major protected by law (under any form of guardianship).
* Lack of informed consent
* Non-beneficiary of the national health insurance system

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Obtention of functional bronchial epithelium from iPSC: yes/no | Day 0 + culture (cross-sectional study)
  Was a functional bronchial epithelium obtained from the patient's induced pluripotent stem cells from blood? (yes/no) The achievement of functional bronchial epithelium (iALI) from iPSCs of a T2 severe asthma patient and an ABPA patient will be assessed by quantification of differentiation markers by immunofluorescence, integrity of the bronchial epithelium by measurement of trans-epithelial resistance (TEER), secretory function by measurement of mucin concentrations (CCSP, MUC5AC and MUC5B) and analysis of ciliary beat

SECONDARY OUTCOMES:
Comparison of the transcriptomic profile between iALI and airway epithelial cells | Day 0 + culture (cross-sectional study)
  the transcriptomic profile of iALI from iPSCs of a T2 severe asthma patient and an ABPA patient will be compare to the one of airway epithelial cells from nasal brushing from the same patients
Comparison of the transcriptomic profile between bronchial epithelia generated from severe asthma patients and from healthy subjects | Day 0 + culture (cross-sectional study)
  The transcriptomic profile of iALI from iPSCs of a T2 severe asthma patient and an ABPA patient will be compare to those from healthy subjects
Differentiation of iPSC into mature eosinophils : yes/no | Day 0 + culture (cross-sectional study)
  Characterization of eosinophils obtained from iPSCs of a T2 severe asthma patient and an ABPA patient by the presence of specific markers by flow cytometry, immunohistochemistry and immunofluorescence
Evaluation of immune cell/bronchial epithelium dialogue | Day 0 + culture (cross-sectional study)
  Co culture of the epithelia with iPSC derived eosinophils and the immune cell/bronchial epithelium dialogue in the co-culture of eosinophils with iALI will be evaluated by the activation of eosinophils in contact with the epithelium and by the characterization and study of the phenotype of the exposed epithelium
Obtention of iPSC from peripheral blood sampling : yes/no | Day 0 + culture (cross-sectional study)
  Qualification of blood-derived iPSC lines by morphology, culture behavior, karyotype and expression of specific markers

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie GAMEZ, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- university Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data will be made available to persons who address a reasonable request to the study director.
  Individual participant data (and an accompanying data dictionary) will be deidentified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
Supporting Information: Study Protocol
Time Frame: Datasets that underlie the results reported in the article (text, tables, figures, and appendices) can be requested after the publication process has been completed.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/ teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.